CLINICAL TRIAL: NCT03123081
Title: Role of Umbilical Cord Milking in the Management of Hypoxic-ischemic Encephalopathy in Neonates: a Randomized Controlled Trial
Brief Title: Role of Umbilical Cord Milking in the Management of Hypoxic-ischemic Encephalopathy in Neonates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Manoj Varanattu, Professor, Department of Neonatology, Jubilee Mission Medical College and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: JubileeMMCRI
Record Dates: First submitted 2017-03-01; First posted 2017-04-21 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blind (Subject)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Umbilical Cord Milking (Experimental): Umbilical Cord Milking involves milking 30 cm length of cord at birth, after initiation of ventilation.
  Interventions: Procedure: Umbilical Cord Milking
- Immediate Umbilical Cord Clamping (No Intervention): Procedure: No Intervention: Immediate Umbilical Cord Clamping or Immediate Cord Clamping.

INTERVENTIONS:
Procedure: Umbilical Cord Milking — At birth the cord of a depressed newborn is clamped immediately and cut 30 cm from the umbilicus. After completion of initial steps, if required, positive pressure ventilation (PPV) is given for 30 seconds, along with UCM. The cord is untwisted and held in a vertical position. It is milked 3 times towards the baby at a speed of 10 cm/s and then clamped 3 cm from the umbilicus. After completion of PPV along with UCM, if the baby requires further resuscitation, the NRP 2015 guidelines will be followed. Depressed newborns who respond to initial steps of resuscitation with normal breathing and heart rate of 100 bpm or higher, will receive UCM after this.
  Other Names: UCM; Umbilical cord stripping
  Arms: Umbilical Cord Milking

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of umbilical cord milking in depressed neonates at birth for prevention of hypoxic ischemic encephalopathy.

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) is a brain injury caused by inadequate supply of oxygen and blood to the brain of a newborn baby. Therapeutic hypothermia is the only proven therapy for these infants. Even after receiving therapeutic hypothermia, 50% of all infants with moderate and severe HIE die or develop neurological and functional impairment. There is a need for a new intervention for neonatal HIE, which is readily available in developing countries and can complement hypothermia.

The American College of Obstetricians and Gynecologists and American Academy of Pediatrics recommend a delay in umbilical cord clamping in vigorous term and preterm infants for at least 30-60 seconds after birth. Immediate umbilical cord clamping is contraindicated in maternal hemodynamic instability, need for immediate resuscitation of the newborn and in conditions where placental circulation is not intact. Umbilical cord milking (UCM) is a simple method of delivering volume and possibly stem cells to those neonates, where resuscitation cannot be postponed for obtaining the benefits of delayed cord clamping.

We hypothesize that depressed neonates who receive umbilical cord milking will have lower incidence and severity of hypoxic ischemic encephalopathy compared to depressed neonates who receive immediate cord clamping.We propose to investigate the safety and effectiveness of UCM in term and late preterm (≥35 week's gestation) infants who are depressed at birth, in preventing the development and/or progression of hypoxic ischemic encephalopathy. The need for immediate resuscitation measures, abnormal parameters (clinical, hematological and biochemical) and neuroimaging will be compared in depressed neonates with and without UCM. If UCM is found to be safe and beneficial, it can be a useful substitute for delayed cord clamping in depressed neonates worldwide.

Conditions: Depressed neonate, Hypoxic-ischemic encephalopathy Intervention: Umbilical cord milking

Study Design Study Type: Interventional Study Design: Allocation: Randomized Endpoint Classification: Efficacy/Safety Study Intervention Model: Parallel Assignment Number of Arms: 2 Masking: Single Blind (Subject) Primary Purpose: Prevention Enrollment: 400 [Anticipated]

Arms and Interventions:

Arms:2, Assigned Interventions: 1. Experimental: Umbilical Cord Milking and 2. No Intervention: Immediate Umbilical Cord Clamping

1. Experimental: Umbilical Cord Milking,Other Name: Umbilical cord stripping Umbilical Cord Milking involves milking a 30 cm long segment of umbilical cord at birth, after initiation of ventilation Procedure: Umbilical Cord Milking (UCM) At birth the umbilical cord of a depressed newborn is clamped immediately and cut 30 cm from the umbilicus and the neonate placed on the resuscitation table. After completion of initial steps, if the baby does not have adequate spontaneous respirations and a heart rate of 100 bpm or higher, positive pressure ventilation (PPV) is given for 30 seconds, along with UCM. The cord is untwisted and held in a vertical position. It is milked 3 times towards the baby at a speed of 10 cm/s and then clamped 3 cm from the umbilicus. The time of cord clamping will be recorded using a timer. After completion of PPV along with UCM, if the baby requires further resuscitation, the NRP 2015 guidelines will be followed. Depressed newborns who respond to initial steps of resuscitation with normal breathing and heart rate of 100 bpm or higher, will receive UCM after this.
2. No Intervention: Immediate Umbilical Cord Clamping, Other Name: routine clamping of the umbilical cord Procedure: Immediate Cord Clamping, At birth the umbilical cord of a depressed newborn is clamped immediately (current recommendation) and cut 3 cm from the umbilicus and the neonate placed on the resuscitation table. The time of cord clamping will be recorded using a timer. After completion of initial steps, if the baby requires further resuscitation, the NRP 2015 guidelines will be followed.

ELIGIBILITY:
Inclusion Criteria:

• Neonates of ≥35 week's gestation and born depressed (defined by NRP 2015 criteria: as those neonates who doesn't cry or breathe at birth and whose tone is poor) in the hospital

Exclusion Criteria:

* MCDA Twin pregnancy (DCDA twins are included)
* Triplet or quadruplet pregnancy
* Presence of IUGR in antenatal scans (< 10th Centile)
* Short umbilical cord length (<30 cm)
* Rh-negative or retrovirus positive mothers
* Major chromosomal or congenital anomalies
* Hydrops fetalis
* Severe placental abruption
* Cord prolapse and cord abnormalities such as true knots
* Culture positive early onset neonatal sepsis

Ages: 1 Minute to 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of HIE in depressed neonates with and without umbilical cord milking | 72 hours
  The severity of HIE if any will be assessed by modified Sarnat staging which is based on level of consciousness, spontaneous activity, neuromuscular control, primitive reflexes, autonomic function and seizures.
  [Designated as safety issue: No];
  Ref:Sarnat HB, Sarnat MS. Neonatal encephalopathy following fetal distress. A clinical and electroencephalographic study. Arch Neurol. 1976; 33:696-705. PMID: 987769

SECONDARY OUTCOMES:
The resuscitation interventions required and the short term outcomes for depressed newborns with and without umbilical cord milking. | 20 minutes after delivery
  The resuscitation interventions required (use of CPAP, oxygen, mask and bag ventilation, endotracheal intubation and ventilation, chest compressions, drugs, and fluid boluses) and the short term outcomes of resuscitation will be assessed using the validated Combined Apgar score (consisting of the Expanded and Specified Apgar scoring systems) introduced by Rudiger et al, in depressed neonates with and without UCM.
  [Designated as safety issue: No];
  Ref:Dalili H, Nili F, Sheikh M, Hardani AK, Shariat M, Nayeri F (2015) Comparison of the Four Proposed Apgar Scoring Systems in the Assessment of Birth Asphyxia and Adverse Early Neurologic Outcomes. PLoS ONE 10(3): e0122116
Requirement of Neonatal Intensive Care Unit (NICU) admission | 1st 24 hours after delivery
  Requirement of Neonatal Intensive Care Unit (NICU) admission [Designated as safety issue: No]
Blood lactate at 24 hours | 1st 24 hours after delivery
  Lactate in the peripheral blood at 24 hours after birth in neonates with any grade of HIE.
  [Designated as safety issue: No]
CD34+ stem cell count at 24 hours | 24 hours after birth
  CD34+ stem cell count in the peripheral blood at 24 hours after birth in neonates with any grade of HIE.
  [Designated as safety issue: No]
The number of neonates with symptomatic polycythemia | 48 hours after birth
  The number of neonates with symptomatic polycythemia defined as lethargy, plethora, jitteriness, tachycardia, tachypnea and with venous hematocrit > 65%.
  [Designated as safety issue: No];
The number of neonates with hyperbilirubinemia requiring phototherapy or exchange transfusion. | 72 hours after birth
  Neonates requiring phototherapy or exchange transfusion will be evaluated according to the NICE/AAP guidelines and serum bilirubin levels will be interpreted according to the baby's age in hours. Physicians who assess the neonate and advice phototherapy or exchange transfusion will be blinded to the intervention.
  [Designated as safety issue: No]
The number of neonates with anemia | 2 hours after birth
  The number of neonates with anemia defined as venous hemoglobin < 12.5 g/dL [Designated as safety issue: No];
MRI changes in the brain of neonates with moderate and severe degrees of HIE who underwent whole body hypothermia. | 14 days after birth
  MRI examination will be performed in neonates who underwent whole body hypothermia 7-14 days after birth and the changes in brain scored as per a validated MR scoring system (Barkovich et al, Am J Neuroradiol 1998;19:143-9) by a neuroradiologist blinded to the intervention.
  [Designated as safety issue: No];
  Ref:Barkovich AJ, Hajnal BL, Vigneron D, Sola A, Partridge JC, Allen F, et al. Prediction of neuromotor outcome in perinatal asphyxia: evaluation of MR scoring systems. Am J Neuroradiol 1998;19:143-9. [PubMed: 9432172]
Duration of hospital stay in neonates with any grade of HIE. | Duration of hospital stay, an expected average of 7-14 days
  Duration of hospital stay in neonates with any grade of HIE. [Designated as safety issue: No]
Survival at 6 weeks of age | 6 weeks after birth
  Survival at 6 weeks of age [Designated as safety issue: No]
Haemoglobin levels at 6 weeks of age | 6 weeks after birth
  Haemoglobin levels at 6 weeks of age [Designated as safety issue: No]
Serum ferritin levels at 6 weeks of age | 6 weeks after birth
  Serum ferritin levels at 6 weeks of age [Designated as safety issue: No]

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Varanattu, MD, Principal Investigator — Jubilee Mission Medical College and Research Institute
Locations (1):
- Jubilee Mission Medical College & Research Institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Upadhyay A, Gothwal S, Parihar R, Garg A, Gupta A, Chawla D, Gulati IK. Effect of umbilical cord milking in term and near term infants: randomized control trial. Am J Obstet Gynecol. 2013 Feb;208(2):120.e1-6. doi: 10.1016/j.ajog.2012.10.884. Epub 2012 Oct 31. PMID 23123382
- [Background] Erickson-Owens DA, Mercer JS, Oh W. Umbilical cord milking in term infants delivered by cesarean section: a randomized controlled trial. J Perinatol. 2012 Aug;32(8):580-4. doi: 10.1038/jp.2011.159. Epub 2011 Nov 17. PMID 22094494
- [Background] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Background] Jaiswal P, Upadhyay A, Gothwal S, Singh D, Dubey K, Garg A, Vishnubhatala S. Comparison of two types of intervention to enhance placental redistribution in term infants: randomized control trial. Eur J Pediatr. 2015 Sep;174(9):1159-67. doi: 10.1007/s00431-015-2511-y. Epub 2015 Mar 24. PMID 25800496
- [Background] Mercer JS, Erickson-Owens DA. Is it time to rethink cord management when resuscitation is needed? J Midwifery Womens Health. 2014 Nov-Dec;59(6):635-644. doi: 10.1111/jmwh.12206. Epub 2014 Oct 8. PMID 25297530
- [Background] Hong Huang, Nicholas Eastman, Brandon Schanbacher et al. Impact of Delayed Cord Clamping on Circulating Progenitor Cells in Extremely Premature Infants. E-PAS 2016:3821.208
- [Background] Aridas JD, McDonald CA, Paton MC, Yawno T, Sutherland AE, Nitsos I, Pham Y, Ditchfield M, Fahey MC, Wong F, Malhotra A, Castillo-Melendez M, Bhakoo K, Wallace EM, Jenkin G, Miller SL. Cord blood mononuclear cells prevent neuronal apoptosis in response to perinatal asphyxia in the newborn lamb. J Physiol. 2016 Mar 1;594(5):1421-35. doi: 10.1113/JP271104. Epub 2015 Dec 14. PMID 26527561
- [Background] Sarnat HB, Sarnat MS. Neonatal encephalopathy following fetal distress. A clinical and electroencephalographic study. Arch Neurol. 1976 Oct;33(10):696-705. doi: 10.1001/archneur.1976.00500100030012. PMID 987769
- [Background] Dalili H, Nili F, Sheikh M, Hardani AK, Shariat M, Nayeri F. Comparison of the four proposed Apgar scoring systems in the assessment of birth asphyxia and adverse early neurologic outcomes. PLoS One. 2015 Mar 26;10(3):e0122116. doi: 10.1371/journal.pone.0122116. eCollection 2015. PMID 25811904
- [Background] Barkovich AJ, Hajnal BL, Vigneron D, Sola A, Partridge JC, Allen F, Ferriero DM. Prediction of neuromotor outcome in perinatal asphyxia: evaluation of MR scoring systems. AJNR Am J Neuroradiol. 1998 Jan;19(1):143-9. PMID 9432172